CLINICAL TRIAL: NCT05908539
Title: A Multi-level and Mixed-method Impact Evaluation for the Jockey Club Elders Get Active Fitness Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGA
Record Dates: First submitted 2023-05-31; First posted 2023-06-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Aging Well
Keywords: Aging; Community-dwelling; Exercise; Care model
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Equipment box (general) (Experimental): A box of exercise equipment is distributed to community dwelling older adults.
  Interventions: Behavioral: Equipment box
- Equipment box with briefing (general) (Experimental): A box of exercise equipment is distributed. Verbal briefing of exercise equipment is provided to community dwelling older adults.
  Interventions: Behavioral: Equipment box with briefing
- Group-based exercise (general) (Experimental): A box of exercise equipment is distributed. Verbal briefing of exercise equipment and an 8-week group exercise training program is provided to community dwelling older adults.
  Interventions: Behavioral: Exercise training
- Group-based exercise with behavioral modification (general) (Experimental): A box of exercise equipment is distributed. Verbal briefing of exercise equipment and an 8-week group exercise training program is provided to community dwelling older adults, following by a 6-week behavioral modification.
  Interventions: Behavioral: Exercise training with behavioral modification
- Equipment box (home-bound) (Experimental): A box of exercise equipment is distributed to home-bound community dwelling older adults.
  Interventions: Behavioral: Equipment box
- Equipment box with briefing (home-bound) (Experimental): A box of exercise equipment is distributed. Verbal briefing of exercise equipment is provided to home-bound community dwelling older adults.
  Interventions: Behavioral: Equipment box with briefing
- Home-based exercise with behavioral modification (home-bound) (Experimental): A box of exercise equipment is distributed. Verbal briefing of exercise equipment and an 8-week group exercise training program is provided to home-bound community dwelling older adults, following by a 6-week behavioral modification.
  Interventions: Behavioral: Exercise training with behavioral modification

INTERVENTIONS:
Behavioral: Equipment box — Participants receive a box of exercise equipment containing dumbbell, elastic band, hand cycle machine, and booklet of exercise instruction only.
  Arms: Equipment box (general); Equipment box (home-bound)
Behavioral: Equipment box with briefing — Participants receive a box of exercise equipment containing dumbbell, elastic band, hand cycle machine, and booklet of exercise instruction, and they are given verbal briefing on how to use the equipment.
  Arms: Equipment box with briefing (general); Equipment box with briefing (home-bound)
Behavioral: Exercise training — Participants receive al box of exercise equipment. They attend an 8-week group exercise training program for 1 hour /session and 1 session/ week, and are supervised by a physical fitness training. The exercise program includes a combination of aerobic, resistance, balance and flexibility exercises.
  Arms: Group-based exercise (general)
Behavioral: Exercise training with behavioral modification — Participants receive al box of exercise equipment. They attend an 8-week group exercise training program for 1 hour /session and 1 session/ week, and are supervised by a physical fitness training. The exercise program includes a combination of aerobic, resistance, balance and flexibility exercises. After finishing the exercise training program, a 6-week behavioral modification is provided. Two home visits and four telephone visits are conducted to empower the participants for exercise at home.
  Arms: Group-based exercise with behavioral modification (general); Home-based exercise with behavioral modification (home-bound)

SUMMARY:
The goal of this clinical trial is provide a scientific evaluation on the impact of the Jockey Club Get Fitness Campaign to improve the physical capacity and health condition of the community-dwelling older adults after the COVID-19 pandemic. Participants will take part in any of the four care models:

* a box of exercise equipment
* a box of exercise equipment with verbal briefing
* a box of exercise equipment and engage in the 8-week group-based exercise training
* receive the wonderful box of exercise equipment and engage in the 8-week group-based exercise training together with the 6-week behavioral modification

Participants with greater physical dependency, greater chronic disease burden or lower motivation for social engagement will take part in any of the three care models:

* a box of exercise equipment only
* a box of exercise equipment with verbal briefing
* a box of exercise equipment and engage in the 4-session home-based exercise training, together with the 6-week behavioral modification

DETAILED DESCRIPTION:
This clinical trial is a mixed-method study which uses multi-level design to compare the effects of different program care models on behavioral and health-related outcomes among two different cohort of community-dwelling older adults. Exercise level and self-efficacy, physical capacity, social connectivity, geriatric symptoms, and health status are measured. A total of 1300 participants will be recruited. Outcome evaluation 8 weeks after intervention and 3 months after intervention will be included to allow the detection of immediate and long-term program benefits. In-depth individual and focus-group interviews will be conducted to solicit the participants' experience and perceived benefits of the program.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years
* Resident of public rental house

Exclusion Criteria:

* Any contraindication to exercise training

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Step count | Changes from baseline to 8 weeks after start intervention
  Step count per day measured by a pedometer
Functional mobility score | Changes from baseline to 8 weeks after start intervention
  Score measured by Life Space Assessment questionnaire (range: 0-120), higher score better performance
Exercise self-efficacy score | Changes from baseline to 8 weeks after start intervention
  Score measured by Self-Efficacy for Exercise Scale questionnaire (range 0-90), higher score higher self-efficacy for exercise
Hand grip strength | Changes from baseline to 8 weeks after start intervention
  Hand grip strength measured by hand-held dynamometer in unit of KG
Performance of timed up-and-go test | Changes from baseline to 8 weeks after start intervention
  Measured by timed up-and-go test in unit of second
Mobility limitation score | Changes from baseline to 8 weeks after start intervention
  Measured by Short Physical Performance Battery (range 0-12), higher score better physical performance
Sarcopenia risk score | Changes from baseline to 8 weeks after start intervention
  Measured by Sarcopenia(SARC) questionnaire and calf circumference in unit of cm (range0-20), higher score higher risk of sarcopenia
Frailty risk score | Changes from baseline to 8 weeks after start intervention
  Measured by Edmonton Frail Scale questionnaire (range0-17), higher score more severer frailty
Social connectedness score | Changes from baseline to 8 weeks after start intervention
  Measured by Social Connectedness Scale questionnaire (20-100), higher score stronger social connectedness
Insomnia risk score | Changes from baseline to 8 weeks after start intervention
  Measured by Insomnia Severity Index questionnaire (range0-28), higher score greater severity of insomnia
Mental health score | Changes from baseline to 8 weeks after start intervention
  Measured by Mental Health Inventory questionnaire (range 0-100), higher score better mental health
Fatigue score | Changes from baseline to 8 weeks after start intervention
  Measured by Brief Fatigue Inventory questionnaire (range0-10), higher score greater fatigue
Loneliness score | Changes from baseline to 8 weeks after start intervention
  Measured by UCLA Loneliness Scale questionnaire (range20-80), higher score greater loneliness
Health status self-rated score | Changes from baseline to 8 weeks after start intervention
  Measured by EQ05D-5L questionnaire (range -0.59-1.0), higher score better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung Yu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided